CLINICAL TRIAL: NCT07297537
Title: Validity and Reliability of the Adductor Endurance Test Developed for the Hip Adductor Muscles
Brief Title: Adductor Endurance Test: Validity and Reliability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Ferruh Taşpınar, Prof. Dr., Izmir Democracy University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HAET-VR-35
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Groin Injury; Hip Injuries; Athletic Injuries
Keywords: Hip adductor muscles; Adductor endurance; Sports injuries; Validity; Reliability
MeSH Terms: conditions — Hip Injuries; Athletic Injuries

STUDY DESIGN:
Intervention Model Description: All participants undergo the Hip Adductor Endurance Test and fixed dynamometer (GroinBar) isometric strength test in randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Group (Experimental): Participants perform the Hip Adductor Endurance Test and GroinBar isometric strength test in randomized order.
  Interventions: Other: Hip Adductor Endurance and Strength Testing

INTERVENTIONS:
Other: Hip Adductor Endurance and Strength Testing — Participants will perform the Hip Adductor Endurance Test to assess adductor muscle endurance, followed by isometric maximum force assessment using the fixed dynamometer (GroinBar) . Tests are conducted in randomized order before routine training sessions, after a 5-minute light aerobic warm-up and dynamic stretching

SUMMARY:
Groin and hip injuries are common in team sports-especially soccer, rugby, and ice hockey-and frequently affect male and young athletes. About 14% of all sports injuries involve the groin and hip region, with most related to the adductor muscles. These injuries often increase during congested match periods and may result in athletes missing 1 to 6.9 weeks of training or competition, extending up to 14 weeks when surgery is required. Weakness in the adductor muscles is a key risk factor for groin injuries, and current assessments primarily measure maximal strength using tools such as squeeze tests, sphygmomanometers, or dynamometers. However, muscle endurance-critical because many injuries occur under fatigue-has not been adequately studied, and no validated endurance tests for the hip adductors exist. This study aims to evaluate the validity and reliability of a newly developed hip adductor endurance test for monitoring endurance strength in professional soccer players.

DETAILED DESCRIPTION:
Groin and hip injuries are common in various team sports such as soccer, rugby, and ice hockey, and are particularly prevalent among male athletes and young athletes aged 15-24 . Studies show that approximately 14% of all injuries occur in the groin and hip regions, and 63% of these are directly related to the adductor muscles . Furthermore, these injuries increase during periods when matches are played at frequent intervals. Research conducted by the Union of European Football Associations (UEFA) within the scope of the Champions League has reported an injury rate of 1.1 per 1,000 match hours for this type of injury. A significant consequence of these injuries is that players are unable to participate in training or matches for an average of 1 to 6.9 weeks ; when surgical intervention is required, this period can extend up to 14 weeks . This situation strains the financial resources of clubs and negatively affects the overall performance of the team . Given the importance of these injuries, it is crucial to regularly monitor athletes' health and take protective measures when necessary . Weakness in the adductor muscles is an important risk factor in predicting groin and hip injury risk. Adductor muscle strength measurements are usually performed using the hip adductor squeeze test, which is both accurate and reliable. During the test, a measuring device is placed between the player's knees, and they are asked to squeeze their legs together. Research has shown that decreased adductor muscle strength may indicate a risk of groin pain development in soccer players. Furthermore, it has been reported that previously injured athletes have weaker adductor muscles compared to uninjured athletes before the season. This information has led to the development of new monitoring methods to detect early signs of muscle weakness in athletes throughout the season and to initiate strengthening exercises. Therefore, the availability and development of easily applicable tests to determine muscle strength may be beneficial for coaches and physical therapists in preventive interventions.

Various technologies such as sphygmomanometers, isometric dynamometers, and isokinetic dynamometers are used to measure adductor strength. In these measurements, peak force variables obtained during isometric contraction of the adductor muscles are recorded. However, all of these methods have been developed to assess the maximum muscle strength of the adductor muscles. Since the vast majority of muscle injuries develop after muscle fatigue, assessing the muscles' ability to resist force over a long period of time may be indicative in predicting muscle injuries. However, there are no studies in the scientific literature on tests used to measure muscle endurance, which is the ability of the hip adductor muscles to resist prolonged force.

The aim of this study is to examine the validity and reliability of the hip adductor endurance test, which will be used to measure hip adductor endurance strength in professional soccer players.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 30 years of age
* Being a professional soccer player for at least four years
* Actively participating in training sessions
* Scoring >87.5 points on the hip and groin injury questionnaire (HAGOS) sports subscale

Exclusion Criteria:

* Having any orthopedic injury involving the lower extremities that would prevent participation in training sessions
* Experiencing pain rated four or higher on the numerical pain rating scale during the hip adductor squeeze test and palpation of the adductor muscle tendons.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment | baseline
  Pain felt during the adductor squeeze test and adductor palpation test, which are applied for inclusion/exclusion criteria, will be assessed using the Numerical Pain Rating Scale. The patient will be asked to mark the level of pain they feel on a 10 cm line, and the marked location will then be measured with a ruler and recorded.
Evaluation of Maximum Isometric Muscle Strength of the Hip Adductor Muscles | baseline
  Hip adductor strength of both lower extremities will be assessed simultaneously using the GroinBar fixed dynamometer (VALD Performance, Australia), a highly reliable method (ICC=0.94). Strength will be measured in two positions: short lever arm (hips 60°, knees 90° flexed, force applied at medial knee epicondyles) and long lever arm (hips and knees extended, force applied 5 cm proximal to medial malleoli). Athletes perform three 5-second maximal isometric contractions per position, with 5-10 seconds rest between repetitions and 20-30 seconds between positions. A trial at 80% of maximal effort is allowed before measurement. Verbal encouragement is provided, and the highest values in Newtons (N) for both dominant and non-dominant legs are recorded; strength ratios are subsequently calculated.
Hip Adductor Endurance Test | baseline
  Hip adductor endurance will be assessed using a time-based version of the Copenhagen Adduction Exercise, which elicits high adductor activation. Participants lie on their side, lift their body concentrically, hold the isometric position as long as possible, and lower eccentrically. The test focuses on maintaining correct alignment and endurance duration rather than maximal force, converting the Copenhagen exercise into an endurance assessment protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Taspinar, Prof.Dr., Principal Investigator — Izmir Democracy University; Ayşe Sezgi Kızılırmak Karataş, Pt.PhD, Study Director — Izmir Democracy University; Mesut Buğday, Pt., Study Director — Göztepe Sports Club
Locations (1):
- Izmir Democracy Univercity, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No